CLINICAL TRIAL: NCT04281615
Title: Examining Perceptions and Brand Approaches for the Canadian 24-Hour Movement Guidelines for Adults
Brief Title: Examining Perceptions of the 24-Hr Movement Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Amy Latimer-Cheung, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Amy Latimer-Cheung, PhD, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6027468
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Health Behavior; Self Efficacy
Keywords: Movement Behaviors; Physical Activity; Sedentary Behaviour; Sleep; Knowledge Translation
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Generic Message) (Experimental): Receives promotional materials that feature a generic messaging approach.
  Interventions: Other: Generic Message
- Control (Threshold Message) (No Intervention): Receives promotional materials that use traditional, threshold messages.

INTERVENTIONS:
Other: Generic Message — Exposed to four sets of promotional materials hypothesized to increase perceptions of self-efficacy to meet Guidelines.
  Arms: Intervention (Generic Message)

SUMMARY:
The main objective of the proposed research is to experimentally test and inform the most effective brand attributes that is to be featured in the forthcoming Canadian 24-Hour Movement Guidelines for Adults. Specifically, there are two main objectives. The first objective is to determine the most preferred tagline associated with the new Guidelines among a sample of Canadian adults. The second objective is to experimentally test if this new attribute fosters stronger perceptions of self-efficacy among an adult sample, when compared to previous threshold-based approaches.

ELIGIBILITY:
Inclusion Criteria:

* between 18-64 years
* Canadian

Exclusion Criteria:

* cannot read/write in English
* already self-reported meeting Guideline recommendations for all three behaviours (physical activity, sedentary behaviour, and sleep)
* self-reported medical condition and/or sleep condition that would prevent individual from meeting the Guideline recommendations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 247 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Change in participants self-efficacy to meet Guidelines measured using the Multi-Dimensional Self-efficacy for Exercise Scale (adapted, scale 0-10; 0=not at all confident, 10=extremely confident) following pre and post exposure to promotional materials. | 3 time points: measuring change from baseline, immediately after viewing message, 2-week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Latimer-Cheung, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Health Studies, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No